CLINICAL TRIAL: NCT04107207
Title: Pilot Study to Evaluate Effects of Kombucha as a Hyperglycemic Therapeutic Agent Within Diabetic Human Subjects
Brief Title: Evaluating the Effects of Kombucha as a Hyperglycemic Therapeutic Agent Within Diabetic Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001101
Record Dates: First submitted 2019-09-01; First posted 2019-09-27 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Double blind crossover
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kombucha Intervention (Active Comparator): Either ginger kombucha or placebo ginger water will be given to subjects for weeks 1-4 and then the reciprocal beverage for weeks 6-10.
  Interventions: Dietary Supplement: Ginger Kombucha
- Placebo Intervention (Placebo Comparator): Either ginger kombucha or placebo ginger water will be given to subjects for weeks 1-4 and then the reciprocal beverage for weeks 6-10.
  Interventions: Dietary Supplement: Ginger Water

INTERVENTIONS:
Dietary Supplement: Ginger Kombucha — Craft Ginger Kombucha, a fermented black tea
  Arms: Kombucha Intervention
Dietary Supplement: Ginger Water — Placebo
  Arms: Placebo Intervention

SUMMARY:
This study's primary objective is to determine the ability of Kombucha to impact blood sugar levels in patients with diabetes mellitus type II. The secondary objective is to determine the ability of Kombucha to impact blood pressure, and quality of life measures as measured by uniform questionnaire that includes: gut health, colds, infections, headaches, sleep, anxiety (GAD2), depression (PHQ2), skin health.

ELIGIBILITY:
Inclusion Criteria:

1. S/he is above the age of 18
2. S/he has the ability to read, speak and write English
3. S/he has telephone access
4. S/he is diabetic and willing to check blood sugar levels every day
5. Hb A1c >7%
6. Possesses a glucometer

Exclusion Criteria:

1. Allergy to kombucha ingredients
2. Drinks kombucha regularly (>3time per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Blood Sugar Levels | 10 weeks
  outcome measure: mg/dL

SECONDARY OUTCOMES:
Gut health | 10 weeks
  Worst ever | worse than usual | average | better than usual | best ever
anxiety | 10 weeks
  How often have you been bothered by the following problems? 6.1. Feeling nervous, anxious or on edge Not at all | Several days | More than half the days | Nearly every day
depression | 10 weeks
  How often have you been bothered by the following problems? 6.3. Little interest or pleasure in doing things Not at all | Several days | More than half the days | Nearly every day
skin health | 10 weeks
  4.1. How would you rate your overall skin health? Worst ever | worse than usual | average | better than usual | best ever 5. How often do you experience skin problems such as dry skin, eczema, rashes, or acne? Not at all | Several days | More than half the days | Nearly every day
vulvovaginal health | 10 weeks
  9.1. How would you rate your overall vulvovaginal health? Worst ever | worse than usual | average | better than usual | best ever

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University MedStar Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mendelson C, Sparkes S, Merenstein DJ, Christensen C, Sharma V, Desale S, Auchtung JM, Kok CR, Hallen-Adams HE, Hutkins R. Kombucha tea as an anti-hyperglycemic agent in humans with diabetes - a randomized controlled pilot investigation. Front Nutr. 2023 Aug 1;10:1190248. doi: 10.3389/fnut.2023.1190248. eCollection 2023. PMID 37588049